CLINICAL TRIAL: NCT01108575
Title: Inspiratory Muscle Strength Training in Ventilator Dependent Patients
Brief Title: Effect of Inspiratory Muscle Training on Duration of Mechanical Ventilation Support
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UF IRB #723-2009
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Respiratory Failure
Keywords: Mechanical ventilation; mechanical ventilation weaning; inspiratory muscle strength training; Patients admitted to a surgical intensive care unit who are expected to receive mechanical ventilation for more than three days.
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory muscle strength training (Experimental)
  Interventions: Other: IMST
- Sham Inspiratory muscle strength training (Sham Comparator)
  Interventions: Other: Sham IMST

INTERVENTIONS:
Other: IMST — inspiratory muscle strength training
  Arms: Inspiratory muscle strength training
Other: Sham IMST — sham inspiratory muscle strength training
  Arms: Sham Inspiratory muscle strength training

SUMMARY:
A growing body of knowledge has documented that the diaphragm, the primary muscle of breathing, atrophies and weakens within days of instituting mechanical ventilation support. Diaphragm weakness has been implicated as a major contributor to difficulty with weaning, or breathing without ventilator support. This study will test whether instituting a diaphragm strength training rehabilitation program will reduce the time patients require mechanical ventilation in a surgical intensive care setting.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to general surgical intensive care unit with respiratory failure and expected to require mechanical ventilation support for more than 72 hours.

Exclusion Criteria:

1. inability to follow simple, one step commands such as "inspire forcefully",
2. patients with prior arrangements to be transferred to other facilities when stabilized,
3. any contraindications to disconnecting pt from ventilator for SHAM or IMST treatment,
4. unstable or difficult airway upon ICU admission and predicted to last for more than 72 hours,
5. use of more than minimal vasopressor or vasodilatatory agents as a continuous infusion,
6. severe dysrhythmias,
7. acute coronary syndrome
8. pulmonary contraindications (pneumon/hemothorax, flail chest),
9. acute surgical problems arising in the immediate post operative period (serious postoperative bleeding, wound dehiscence, etc). When and if these problems resolve and the patient meets other entry criteria, they will be eligible to be recruited for participation.
10. active neuromuscular diseases that would prevent or interfere with responding to strength training (e.g., amyotrophic lateral sclerosis, multiple sclerosis, myasthenia gravis, polymyositis, muscular dystrophy or other dystrophies and myopathies)
11. spinal cord injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation support | Patients will be observed for up to 28 days following admission to the ICU

SECONDARY OUTCOMES:
Maximal inspiratory pressure | Patients will be observed for up to 28 days following admission to the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States